CLINICAL TRIAL: NCT02158650
Title: The Efficiency and Effectiveness of Using Video-Based Treatment Option Education Medium for Basal Cell Carcinoma Patients
Brief Title: Video-Based Treatment Options for Basal Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Suephy Chen, MD, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00058881; DCOR-BCC (Other: Other); IRB00074984 (VA IRB number) (Other: Other)
Record Dates: First submitted 2014-06-02; First posted 2014-06-09 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Basal Cell Carcinoma
Keywords: informed consent; video-based
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video Group (Experimental): Patients randomized to Group II will be emailed the educational video, pre- and post- knowledge assessments, and patient satisfaction survey with instructions on what order to fill them out. Group II patients will report to the treatment visit and undergo discussion of options and treatment as per standard of care. An additional knowledge assessment survey will be administered to Group II patients after discussion with treating physician.
  Interventions: Behavioral: Video-Based Informed Consent
- Control Group (No Intervention): Patients randomized to Group I will be come to the clinic for the treatment visit and discuss options and treatment as per standard of care. Pre- and post- discussion knowledge assessments and satisfaction surveys will be administered at the time of the treatment visit.

INTERVENTIONS:
Behavioral: Video-Based Informed Consent
  Arms: Video Group

SUMMARY:
The purpose of this study is to determine if presenting treatment options to basal cell carcinoma patients in video format will improve efficiency and allow patients to receive consistent, comprehensive, visually-depicted treatment option information to improve patient quality of care. Patients can learn more about treatment options as they are depicted visually so as to better assist them in understanding treatment risks and benefits to confidently make a well-informed decision. Primarily, the study will evaluate efficiency when using the education video medium. The study will also evaluate the effectiveness of the video medium as an aid to decision making in addition to standard of care in comparison to the standard of care alone. Additionally, the study will evaluate both patients' and dermatologists' satisfaction of the educational intervention.

DETAILED DESCRIPTION:
Currently, verbal consultation is the widespread practice in presenting treatment options for basal cell carcinoma patients. This method, although personable and direct, is often incomplete and subject to variability.

The Emory Department of Dermatology has created an educational video involving treatment options for patients with newly diagnosed basal cell carcinoma as part of routine clinical care. The purpose of this study is to determine the effectiveness of the video format in improving efficiency and workflow. Many studies have shown that multimedia tools improve patient education and have been more efficient than in-office verbal discussions alone. In addition, educational videos have been documented to increase patient satisfaction as well as decrease patient stress level and anxiety. Other advantages of educational videos are for the repetition and reinforcement that would benefit the patient.

Moreover, with the utilization of video, patients will receive the same comprehensive information, making the delivery reproducible and controlled. With verbal communication, there is usually no standardized interaction between staff and patients to ensure that the patient is receiving all pertinent information regarding their options. For example, a study designed to examine retention rates for verbal and written instructions, including 10 potential complications, in patients undergoing Mohs micrographic surgery showed an overall poor retention rate of only 26.5% just 20 minutes after being informed. It is obvious then that educational protocols need additional modalities in order to improve overall retention rates. This then suggests that information presented in video format increases knowledge retention in patients, even weeks after initial delivery of information.

Study participants will be randomly assigned to the control (Group I) - or video- (Group II) group. Participants will be randomized by clinic. Patients randomized to Group II will complete a pre-video knowledge assessment followed by viewing of the BCC educational video. Patients will complete a post-video knowledge assessment following video viewing. Group II patients will then undergo discussion of treatment options with their physician as per standard of care. After the treatment discussion, Group II patients will complete an additional knowledge assessment. After the treatment visit is complete, patients will complete a satisfaction survey. Patients randomized to Group I will not view the educational video. Group I patients will complete a pre-knowledge assessment before their standard of care discussion of treatment options with their physician. Similar to Group II, patients in Group I complete an additional knowledge assessment after the treatment discussion and a satisfaction survey at the conclusion of the treatment visit.

If there is failure of completion of a satisfaction survey in the dermatology clinic, patients (group I and group II) may be contacted via phone to complete the survey.

Physicians will be recruited to complete a satisfaction survey at the end of the day only if they provided treatment to a Group II patient (patients who viewed the video).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed basal cell carcinoma (BCC) patients aged 18 or above for which treatment of Mohs surgery is not necessary and who agree to voluntarily participate in the study

Exclusion Criteria:

* Newly diagnosed basal cell carcinoma patients with an aggressive histologic subtype of BCC or for which treatment by Mohs surgery is deemed necessary based on clinician assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | Up to 1 hour (end of clinic visit)
  Paper surveys

SECONDARY OUTCOMES:
Physicians' satisfaction | Up to 10 hours (end of clinic day)
  Online satisfaction survey
Change in health knowledge | Baseline (beginning of clinic visit), up to 1 hour (end of clinic visit)
  Paper surveys
Video Medium Effectiveness | Baseline (beginning of clinic visit), up to 1 hour (end of clinic visit)
  Paper surveys

CONTACTS AND LOCATIONS:
Overall Officials: Suephy Chen, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia

REFERENCES:
- [Background] Armstrong AW, Alikhan A, Cheng LS, Schupp C, Kurlinkus C, Eisen DB. Portable video media for presenting informed consent and wound care instructions for skin biopsies: a randomized controlled trial. Br J Dermatol. 2010 Nov;163(5):1014-9. doi: 10.1111/j.1365-2133.2010.10067.x. PMID 20977443
- [Background] Eggers C, Obliers R, Koerfer A, Thomas W, Koehle K, Hoelscher AH, Bollschweiler E. A multimedia tool for the informed consent of patients prior to gastric banding. Obesity (Silver Spring). 2007 Nov;15(11):2866-73. doi: 10.1038/oby.2007.340. PMID 18070779
- [Background] Fleischman M, Garcia C. Informed consent in dermatologic surgery. Dermatol Surg. 2003 Sep;29(9):952-5; discussion 955. doi: 10.1046/j.1524-4725.2003.29251.x. PMID 12930338
- [Background] Migden M, Chavez-Frazier A, Nguyen T. The use of high definition video modules for delivery of informed consent and wound care education in the Mohs Surgery Unit. Semin Cutan Med Surg. 2008 Mar;27(1):89-93. doi: 10.1016/j.sder.2008.02.001. PMID 18486030
- [Background] Schenker Y, Fernandez A, Sudore R, Schillinger D. Interventions to improve patient comprehension in informed consent for medical and surgical procedures: a systematic review. Med Decis Making. 2011 Jan-Feb;31(1):151-73. doi: 10.1177/0272989X10364247. Epub 2010 Mar 31. PMID 20357225
- [Background] Shukla AN, Daly MK, Legutko P. Informed consent for cataract surgery: patient understanding of verbal, written, and videotaped information. J Cataract Refract Surg. 2012 Jan;38(1):80-4. doi: 10.1016/j.jcrs.2011.07.030. Epub 2011 Nov 6. PMID 22062774
- [Background] Weston J, Hannah M, Downes J. Evaluating the benefits of a patient information video during the informed consent process. Patient Educ Couns. 1997 Mar;30(3):239-45. doi: 10.1016/s0738-3991(96)00968-8. PMID 9104380